CLINICAL TRIAL: NCT03915366
Title: Empirical Treatment Against Cytomegalovirus and Tuberculosis in HIV-infected Infants With Severe Pneumonia: a Multicenter, Open-label Randomized Controlled Clinical Trial
Brief Title: Empirical Treatment Against Cytomegalovirus and Tuberculosis in HIV-infected Infants With Severe Pneumonia
Acronym: EMPIRICAL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: University Hospital, Bordeaux (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); PENTA Foundation (Network); Centre Hospitalier Cocody (Unknown); Malawi-Liverpool-Wellcome Trust Clinical Research Programme (Other); Eduardo Mondlane University (Other); Centro de Investigação em Saúde de Manhiça (Other); Stichting Katholieke Universiteit (Other); Barcelona Institute for Global Health (Other); University of Lincoln (Other); Makerere University (Other); University Teaching Hospital, Lusaka, Zambia (Other); University of Zimbabwe (Other); Kamuzu Central Hospital (Other); Servicio Madrileño de Salud, Madrid, Spain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19/096; 2019-001749-42 (EudraCT Number); EDCTP RIA2017MC-2013EMPIRICAL (Other Grant/Funding Number: EDCTP); U1111-1231-4736 (Other: Universal Trial Number); PACTR201904797961340 (Other: Pan African Clinical Trial Registry)
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Pneumonia; HIV/AIDS; Tuberculosis; Cytomegalovirus Infections
MeSH Terms: conditions — Pneumonia; Acquired Immunodeficiency Syndrome; Tuberculosis; Cytomegalovirus Infections | interventions — Valganciclovir; Therapeutics; Antitubercular Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of Care (SoC) (No Intervention): Standard treatment for severe pneumonia and pneumonia in HIV-infected infants:
  Ceftriaxone 80 mg/k/day or Ampicillin plus Gentamicin ampicillin 50 mg/kg, or benzylpenicillin 50,000 unit/kg im/iv every six hours plus Gentamicin 7.5 mg/kg/im or iv once a day Cotrimoxazole trimethoprim (TMP) 8mg/kg/dose + sulfamethoxazole (SMX) 40mg/kg/dose three times daily Prednisolone 2mg/kg during 7 days, plus 1mg/kg other 7 days, plus 0.5 mg/kg for 7 days
- Valganciclovir plus SoC (Experimental): Treatment for cytomegalovirus (CMV) Valganciclovir (powder for suspension, 50 mg/mL) oral, 16 mg/kg/12 hours for 15 days, and Standard or Care as described in Control Group
  Interventions: Drug: Valganciclovir Oral Solution [Valcyte]
- Tuberculosis Treatment plus SoC (Experimental): Treatment for tuberculosis Fixed-dose dispersible tablet of rifampicin, isoniazid, pyrazinamide (75/50/150 mg) Fixed-dose dispersible tablet of rifampicin/isoniazid (75/50 mg) Ethambutol 100 mg dispersible tablet Plus Standard of Care described in the Control Group
  Doses of tuberculosis treatment:
  Isoniazid 10 mg/kg (range 7-15 mg/kg)/day; maximum dose 300 mg/day for 6 months.
  Rifampicin 15 mg/kg (range 10-20 mg/kg)/day; maximum dose 600 mg/day for 6 months.
  Pyrazinamide 35 mg/kg (range 30-40 mg/kg)/day for 2 months. Ethambutol 20 mg/kg (range 15-25 mg/kg)/day for 2 months.
  Interventions: Drug: Tuberculostatic Agents
- Tuberculosis Treatment plus Valganciclovir plus SoC (Experimental): Treatment for CMV and for tuberculosis. Fixed-dose dispersible tablet of rifampicin, isoniazid, pyrazinamide (75/50/150 mg) Fixed-dose dispersible tablet of rifampicin/isoniazid (75/50 mg) Ethambutol 100 mg dispersible tablet Valganciclovir (powder for suspension, 50 mg/mL) oral, 16 mg/kg/12 hours for 15 days, Plus Standard of Care described in the Control Group
  Doses of tuberculosis treatment:
  Isoniazid 10 mg/kg (range 7-15 mg/kg)/day; maximum dose 300 mg/day for 6 months.
  Rifampicin 15 mg/kg (range 10-20 mg/kg)/day; maximum dose 600 mg/day for 6 months.
  Pyrazinamide 35 mg/kg (range 30-40 mg/kg)/day for 2 months. Ethambutol 20 mg/kg (range 15-25 mg/kg)/day for 2 months.
  Interventions: Drug: Valganciclovir Oral Solution [Valcyte]; Drug: Tuberculostatic Agents

INTERVENTIONS:
Drug: Valganciclovir Oral Solution [Valcyte] — Treatment for CMV
  Other Names: Treatment for CMV
  Arms: Tuberculosis Treatment plus Valganciclovir plus SoC; Valganciclovir plus SoC
Drug: Tuberculostatic Agents — Treatment for tuberculosis
  Other Names: Treatment for TB
  Arms: Tuberculosis Treatment plus SoC; Tuberculosis Treatment plus Valganciclovir plus SoC

SUMMARY:
This trial will evaluate whether empirical treatment against cytomegalovirus and tuberculosis improves survival of HIV-infected infants with severe pneumonia.

DETAILED DESCRIPTION:
Pneumonia is the main cause of death in Human Immunodeficiency Virus (HIV)-infected children. A significant number of undiagnosed or poorly treated HIV-infected children present to health services with severe pneumonia. World Health Organization (WHO) guidelines to treat severe pneumonia in HIV-infected infants include empirical treatment against common bacteria plus Pneumocystis jirovecii. Although this approach has contributed to reducing overall case fatality rates, mortality in this particularly vulnerable group remains unacceptably high. Autopsy studies in Africa have shown that cytomegalovirus (CMV) infection and tuberculosis (TB) are important underdiagnosed and undertreated causes of deaths. Our objective is to evaluate whether empirical treatment against cytomegalovirus and tuberculosis improves survival of HIV-infected infants with severe pneumonia. A randomized factorial clinical trial will be conducted in six sub-Saharan African countries to evaluate the safety and efficacy of empirical treatment against cytomegalovirus and tuberculosis in HIV-infected infants aged 28 days to 365 days admitted to hospital with severe pneumonia. The primary outcome is mortality. All HIV-infected infants will receive standard of care (SoC) pneumonia treatment, including antibiotics, cotrimoxazole, and prednisolone. A group of patients will receive SoC, another group will receive valganciclovir plus SoC, another group will receive tuberculosis treatment plus SoC, and another group will receive valganciclovir, tuberculosis treatment, and SoC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 28 days to 365 days of age
2. Pneumonia defined as chest indrawing or fast breathing for age, for infants 28 to 60 days of age ≥60 breaths per minute and for infants 61 to 365 days of age, ≥50 breaths per minute.
3. Current hospitalization due to pneumonia with criteria for parenteral antibiotics (1 or more criteria)

   1. Chest indrawing with HIV infection
   2. No improvement with oral treatment.
   3. One or more danger signs according to WHO 5,44,45

      * Central cyanosis or saturation of O2 <90%
      * Severe respiratory distress, e.g. grunting or very severe chest indrawing
      * Signs of pneumonia with a general danger sign:
      * Unable to drink or breastfeed
      * Persisting vomiting
      * Convulsions in the last 24 hours
      * Lethargic or unconscious
      * Stridor while calm
      * Severe malnutrition
4. HIV-confirmed infection (with at least one molecular method: DNA polymerase chain reaction (PCR) or RNA PCR/viral load).
5. Informed consent obtained

Exclusion Criteria:

1. Clinical TB (pulmonary or extrapulmonary) diagnosis, defined as the necessity of TB-T prescribed by a physician, at the moment of randomization
2. Known bacteriologically confirmed TB case (at least one biological specimen positive by culture or Xpert MTB/RIF) at the moment of randomization
3. Patient previously treated for TB or currently on treatment for TB
4. Documented evidence of close TB exposure (household contact of a patient with documented TB during the lifetime of the child, or currently receiving TB-T)
5. Pure wheezers defined as a clear clinical improvement after a bronchodilator test (give a challenge of rapid-acting inhaled bronchodilator for up to three times 15-20 minutes apart. Count the breaths and look for chest indrawing again, and then re-classify)
6. Active malignancies
7. Systemic immunosuppressive medications. Steroids will be considered to be immunosuppressing only if >2 mg/kg of prednisone or equivalent during >15 days
8. Evidence of condition other than HIV and pneumonia which precludes, to the judgment of the clinical researcher, enrollment in this trial due to risk for the patient. In case of doubt, the Trial Management Team will be contacted to assess eligibility
9. Less than 2.5 kg of weight
10. Hb <6 g/dL in the screening blood test or in a test done in the last 48 hours. Transfusion is permitted to achieve >6 g/dL if the patient's state allows it. In case a transfusion is administered, the patient can be enrolled
11. Neutropenia <500 /mm3 in the screening blood test or in a test done in the last 48 hours. Repeating the test is allowed to check eligibility

Ages: 28 Days to 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 563 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  The primary endpoint of the study is all-cause mortality, focusing on the short term (up to 15-days) and long-term (up to 1-year) mortality. Mortality will be calculated using all-cause mortality after the admission over all the trial time.

SECONDARY OUTCOMES:
Days with oxygen therapy | 60 days
  1. Duration of oxygen requirements (in days, from the first requirement until definitive withdrawal, being day 1 the first day of oxygen requirement).
Days of hospitalization | 1 year
  2. Cumulative days of hospitalization from discharge to day +365 after enrollment
Serious Adverse Events | 1 year
  Serious Adverse Events (SAEs), this is, grade 3 and 4 AEs.
Adverse Reactions | 1 year
  Adverse Reactions (AR)
Notable Adverse Events | 1 year
  Adverse events (AEs) requiring stop of investigational medical product (IMP), all AEs relevant for risk/benefit ratio, including infections, liver toxicity, neurological and optic toxicity, renal, hematological and any AE grade 1, 2, 3 or 4 that the investigator estimates to be relevant
Immune-reconstitution inflammatory syndrome | 6 months
  Incidence of TB-related immune-reconstitution inflammatory syndrome (IRIS)
Baseline cytomegalovirus prevalence | 30 days
  Baseline prevalence of CMV infection and CMV-attributable pneumonia (based in a CMV viral load threshold) in recruited HIV-infected infants with severe pneumonia
Baseline tuberculosis prevalence | 60 days
  Baseline prevalence of microbiological confirmed and unconfirmed TB (according to Graham criteria, Updated Clinical Case Definitions for Classification of Intrathoracic Tuberculosis in Children 2015) in recruited HIV-infected patients with severe pneumonia
Tuberculosis incidence | 1 year
  New confirmed and unconfirmed TB cases according to Graham criteria during 1-year of follow-up among patients without TB-T
Deaths attributable to tuberculosis | 1 year
  Proportion of confirmed and unconfirmed TB, according to Graham criteria, in died children
CMV prevalence in died participants | 1 year
  Proportion of CMV infection in died children
CMV Molecular response to treatment | 1 year
  Reduction of quantitative CMV viral load in blood and saliva in infants treated with valganciclovir from enrollment to day +15
TB-lipoarabinomannan (LAM) sensitivity and specificity | 1 year
  To assess the diagnostic accuracy (sensitivity and specificity) of TB-LAM for the diagnosis of confirmed TB (reference: positive Xpert Mycobacterium tuberculosis (MTB)/RIF Ultra in feces and/or NPA)
Quality-adjusted life expectancy | 1 year
  Economic evaluation for quality-adjusted life expectancy
Per-patient cost | 1 year
  Economic evaluation of the treatments (per-patient cost)

CONTACTS AND LOCATIONS:
Overall Officials: Cinta Moraleda, MD, PhD, Study Chair — Fundación para la Investigación Biomédica del Hospital 12 de Octubre
Locations (13):
- Programme PACCI. Centre Hospitalier Cocody., Abidjan, Côte d’Ivoire
- France (2):
  - Université de Bourdeaux, Bourdeaux
  - INSERM, Toulouse
- PENTA Foundation, Padua, Italy
- Malawi Liverpool Welcome Trust. Queen Elizabeth Central Hospital College of Medicine, Blantyre, Malawi
- Mozambique (2):
  - Cemtro de Investigaçao em Saúde da Manhiça, Manhiça
  - Hospital Central Maputo, Maputo
- Stichting Katholieke Universiteit Radboudumc, Nijmegen, Netherlands
- Fundación para la Investigación Biomédica del Hospital 12 de Octubre, Madrid, Spain
- Makerere University - Mulago Hospital, Kampala, Uganda
- University of Lincoln, Lincoln, United Kingdom
- Lusaka Teaching Hospital, Lusaka, Zambia
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes
After principal results, addressing primary and secondary objectives will be published. A final repository will be chosen for anonymized data sharing, and transparency after the trial is closed, according to the funder (EDCTP) rules and recommendations, unless national laws impede it.
Time Frame: Within 12 months of the completion of the study.
Access Criteria: The repository will be public-available by concrete permission of the Clinical Trial Unit. Those interested in having the database or any of its subsets should provide concrete research proposal that may be accepted under citation condition.

REFERENCES:
- [Derived] Dominguez-Rodriguez S, Lora D, Tagarro A, Moraleda C, Ballesteros A, Madrid L, Manukyan L, Marcy O, Leroy V, Nardone A, Burger D, Bassat Q, Bates M, Moh R, Tam PI, Mvalo T, Magallhaes J, Buck WC, Sacarlal J, Mussime V, Chabala C, Mujuru HA, Rojo P; EMPIRICAL group. Statistical analysis plan for the "empirical treatment against cytomegalovirus and tuberculosis in HIV-infected infants with severe pneumonia" clinical trial. Trials. 2025 Apr 30;26(1):144. doi: 10.1186/s13063-025-08841-7. PMID 40307889
- [Derived] Jacobs TG, Mumbiro V, Chitsamatanga M, Namuziya N, Passanduca A, Dominguez-Rodriguez S, Tagarro A, Nathoo KJ, Nduna B, Ballesteros A, Madrid L, Mujuru HA, Chabala C, Buck WC, Rojo P, Burger DM, Moraleda C, Colbers A; EMPIRICAL Clinical Trial Group; EMPIRICAL Clinical Trial Group. Brief Report: Suboptimal Lopinavir Exposure in Infants on Rifampicin Treatment Receiving Double-dosed or Semisuperboosted Lopinavir/Ritonavir: Time for a Change. J Acquir Immune Defic Syndr. 2023 May 1;93(1):42-46. doi: 10.1097/QAI.0000000000003168. Epub 2023 Apr 1. PMID 36724434
- [Derived] Rojo P, Moraleda C, Tagarro A, Dominguez-Rodriguez S, Castillo LM, Tato LMP, Lopez AS, Manukyan L, Marcy O, Leroy V, Nardone A, Burger D, Bassat Q, Bates M, Moh R, Iroh Tam PY, Mvalo T, Magallhaes J, Buck WC, Sacarlal J, Musiime V, Chabala C, Mujuru HA. Empirical treatment against cytomegalovirus and tuberculosis in HIV-infected infants with severe pneumonia: study protocol for a multicenter, open-label randomized controlled clinical trial. Trials. 2022 Jun 27;23(1):531. doi: 10.1186/s13063-022-06203-1. PMID 35761406